CLINICAL TRIAL: NCT04225468
Title: Safe Options for ACL Recovery: An Opioid Exposure Reduction Program for Anterior Cruciate Ligament Surgery Patients
Brief Title: Safe Options for ACL Recovery
Acronym: SOAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Derefinko, PhD (Other)
Collaborators: University of Memphis (Other); Campbell Clinic (Other)
Responsible Party: Sponsor-Investigator, Karen Derefinko, PhD, Assistant Professor, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-07075-XP
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Anterior Cruciate Ligament Injuries; Opioid Use
Keywords: prevention; opioid exposure; exposure reduction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment As Usual (TAU) (No Intervention): No intervention will be administered.
- Opioid Exposure Reduction Program 1 (OERP1) (Experimental): Participants will engage in a brief, educational intervention at their pre-surgery appointment approximately 2-3 weeks before ACL reconstruction surgery.
  Interventions: Behavioral: ACL Opioid Exposure Reduction Program
- Opioid Exposure Reduction Program 2 (OERP2) (Experimental): Participants will engage in the same intervention as OERP1, but those in OERP2 will also receive a 5-minute "booster" intervention session 3 days after surgery.
  Interventions: Behavioral: ACL Opioid Exposure Reduction Program

INTERVENTIONS:
Behavioral: ACL Opioid Exposure Reduction Program — Subjects will engage in a brief, educational which includes information about the appropriate use of opioid pain medication, exposure and tolerance, the definition of misuse and opioid-related harms, how to wean off medication, alternative pain management strategies, and appropriate disposal of leftover medication.
  Other Names: ACL-OERP
  Arms: Opioid Exposure Reduction Program 1 (OERP1); Opioid Exposure Reduction Program 2 (OERP2)

SUMMARY:
The purpose of the proposed work is to test a brief opioid exposure reduction program (ACL-OERP) designed to improve health literacy about opioid use following surgeries. This intervention is specifically designed to be used with patients (or for patients under 18, the patient and caregiver) undergoing Anterior Cruciate Ligament (ACL) reconstruction, a painful surgery that is often followed by at least 7 days of opioid medication.

DETAILED DESCRIPTION:
The goal of this study is to test whether the ACL-OERP intervention (vs. a treatment as usual [TAU] comparison) improves knowledge of (1) risks associated with opioid self-administration (development of tolerance, dangers of concomitant sedative use, taking as prescribed for safety), (2) expected pain following ACL reconstruction, (3) accurate pain assessment, (4) and weaning from opioid to non-narcotic analgesics.

There will be one control arm (TAU) and two intervention arms, both of which are experimental. Both will receive the ACL-OERP before surgery, and the second arm will also receive a "booster" intervention session of the intervention 3 days after surgery.

In addition, investigators wish to compare the amount of opioid self-administered in the intervention groups (vs. TAU comparison) to assess whether this knowledge reduces self-administration of opioid. The project will also examine whether the implementation of the booster intervention session in the third arm improves these outcomes compared to the other intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for a pre-operatory appointment at the study site for ACL reconstruction with patellar tendon autograft surgery.
* Be able to return to the clinic at least one time within the first 10 days post-op.

Exclusion Criteria:

* Under 12 years of age
* Contraindication to opioids
* Unable to understand intervention material in English

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Total morphine milligram equivalents administered | Assessed at 30 days post surgery
  Cumulative morphine milligram equivalents self-administered following surgery; based upon pill counts

SECONDARY OUTCOMES:
Knowledge of safe opioid use | Assessed at baseline and 7-days post surgery
  Change in pre and post test scores of a knowledge test of topics covered in the intervention including tolerance, weaning off opioids, safe disposal methods, and alternative pain management strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that a cleaned data set of study-specific data will be provided within two years following the termination of the study for the data archive and this data set would be made public. Confidentiality of individual participants would be maintained with all releases of data. The final study analytical database would be processed according to HIPAA definitions for public data sharing. Documentation would be provided along with the data sharing file that includes but is not limited to: data dictionary, data codebook, valid variable ranges (where provided), the protocol, procedure and operational manuals, intervention manual or programs and any electronic versions of any paper forms that were used in data collection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after data collection ends

REFERENCES:
- See also: UTHSC main website — https://uthsc.edu